CLINICAL TRIAL: NCT00895921
Title: Acute Impact of Antipsychotics on Insulin Sensitivity: A Novel Human Model
Brief Title: Examining the Effects of Antipsychotic Medications on Insulin Sensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jonathan M. Meyer, MD, Research Scientist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R21MH082805 (NIH); R21MH082805 (NIH); DATR A5-ETSE; 071224 (Other: UCSD HRPP (IRB))
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Diabetes
Keywords: Insulin Resistance; Antipsychotic Medications
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Olanzapine; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole (Active Comparator): Participants will receive an injection of aripiprazole during the tracer-clamp study.
  Interventions: Drug: Aripiprazole
- Olanzapine (Active Comparator): Participants will receive an injection of olanzapine during the tracer-clamp study.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Single intramuscular 10-mg dose
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Aripiprazole — Single intramuscular 9.75-mg dose
  Other Names: Abilify
  Arms: Aripiprazole

SUMMARY:
This study will examine the effects of two different antipsychotic medications on control of blood sugar in people who are at risk of diabetes but mentally healthy.

DETAILED DESCRIPTION:
Antipsychotic medications are those that treat the most severe psychiatric symptoms, such as hallucinations, paranoid thoughts, and delusions. Research shows that some of these medications may put people at a higher risk of metabolic derangements, such as insulin resistance. Certain antipsychotics, like clozapine and olanzapine, are associated with a higher risk of metabolic side effects than others, like aripiprazole and ziprasidone. Because people with schizophrenia may experience adverse side effects from switching antipsychotic medications and because it is difficult to find people with schizophrenia who do not have experience taking antipsychotics, this study will use people without psychiatric disorders who are at risk for diabetes in place of people with schizophrenia. The study will compare the effects of single doses of two antipsychotic medications, olanzapine and aripiprazole, on insulin action in this population. In addition to determining metabolic effects of these medications, this study will also seek to demonstrate the feasibility of using mentally healthy people at risk of diabetes as a substitute for people with schizophrenia in studying these effects.

Participation in this study will last 4 weeks. Participants will first complete a screening visit that will include the following: an oral glucose tolerance test (OGTT), which involves a blood draw, consumption of a sugar drink, and then a second blood draw; a review of medical and psychiatric history, including use of medicines and psychiatric medications; and measurement of participants' height and weight. The second visit, scheduled 2 weeks after screening, will include a tracer-clamp study to test how participants' bodies handle sugar. The tracer-clamp study will be conducted over the course of one night and morning and will require participants to stay at the study location overnight. At 3 AM, participants will receive an intravenous line (IV) with a sugar solution. Just before 8 AM, they will receive a second IV in the opposite arm that will draw blood and monitor blood sugar levels.

At 8 AM, participants will begin receiving insulin in the first IV; blood samples will be drawn and blood sugar levels will be monitored during this time to ensure they remain within a healthy range. At 11 AM, participants will receive an injection of an antipsychotic medication into their arm muscles. The antipsychotic, which will be randomly assigned, will be either olanzapine or aripiprazole. Participants will be monitored for 3 hours after receiving the injection of antipsychotic medication; during this time, more blood samples will be drawn, blood sugar levels will be monitored to ensure they are within a healthy range, and secondary medications will be available to counteract certain side effects of the antipsychotics. After 2 more weeks, participants will undergo a third study visit in which they repeat the OGTT.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetic, defined as 2-hour post-load serum glucose between 140 and 199 mg/dl on a 75-gram standard oral glucose tolerance test (OGTT) within the past 90 days
* Family history of type 2 diabetes mellitus
* Body mass index (BMI) between 25 and 35 kg/m2
* English speaker
* Nonsmoker

Exclusion Criteria:

* History of Axis I mood, anxiety, or psychotic disorder, confirmed by Structured Clinical Interview for DSM-IV
* Use of psychotropic drugs

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M. Meyer, MD, Principal Investigator — UCSD and Veterans Affairs San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Participants will receive an injection of aripiprazole during the trace-clamp study.
  Aripiprazole: Single intramuscular 9.75-mg dose
- Olanzapine: Participants will receive an injection of olanzapine during the trace-clamp study.
  Olanzapine: Single intramuscular 10-mg dose
Period: Overall Study
Arm/Group | Aripiprazole | Olanzapine
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Male subjects ages 40-65 with impaired glucose tolerance as measured by oral glucose tolerance testing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Olanzapine | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (5.57) | 54.4 (5.97) | 51.17 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Glucose Disposition [Mean (Standard Deviation); unit: mg/kg/min] — Glucose disposition is measured using the hyperglycemic clamp technique. This method allows one to measure either how well an individual metabolizes glucose or how sensitive an individual is to insulin.
  mg/kg/min | 3.88 (1.99) | 3.31 (1.35) | 3.60 (1.67)
Insulin Suppression of Endogenous Glucose Production (EGP) [Mean (Standard Deviation); unit: % suppression of EGP] | 84.28 (20.30) | 86.52 (22.34) | 85.40 (21.32)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glucose Disposition
Description: Ratio of post-antipsychotic/pre-antipsychotic glucose disposition as measured using the hyperglycemic clamp technique. This method allows one to measure either how well an individual metabolizes glucose or how sensitive an individual is to insulin.
Time Frame: Measured over 6 hours
Measure: Mean (Standard Deviation); unit: ratio of post/pre values
Arm/Group | Aripiprazole | Olanzapine
Number analyzed (Participants) | 15 | 15
ratio of post/pre values | 1.18 (.324) | 1.42 (.300)
Statistical Analysis 1: Comparison: Aripiprazole vs Olanzapine; Test type: Superiority or Other; p = 0.042, t-test, 2 sided — The a priori threshold for statistical significance is <0.05; Mean Difference (Final Values) = .242, 95% CI 2-sided [.00943 to .47605], Standard Error of Mean .1139

2. Secondary Outcome: Change in Percent of Insulin Suppression of Endogenous Glucose Production
Description: Ratio of Post-Antipsychotic/Pre-Antipsychotic Percent of Insulin Suppression of Endogenous Glucose Production
Time Frame: Measured over 6 hours
Measure: Mean (Standard Deviation); unit: ratio of post/pre values
Arm/Group | Aripiprazole | Olanzapine
Number analyzed (Participants) | 15 | 15
ratio of post/pre values | 1.0594 (.519) | 1.312 (.642)
Statistical Analysis 1: Comparison: Aripiprazole vs Olanzapine; Test type: Superiority or Other; p = 0.269, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05; Mean Difference (Final Values) = .253, 95% CI 2-sided [-0.208 to 0.714], Standard Error of Mean 0.224

3. Secondary Outcome: Akathisia
Description: Number of subjects reporting mild or greater complaints of akathisia after antipsychotic administration
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Aripiprazole | Olanzapine
Number analyzed (Participants) | 15 | 15
participants | 1 | 7
Statistical Analysis 1: Comparison: Aripiprazole vs Olanzapine; Comparison of akathisia rates between the two arms; Test type: Superiority or Other; p = 0.012, Chi-squared, Corrected; Mean Difference (Net) = 0.400, 95% CI 2-sided [.095 to .705], Standard Error of Mean 0.149

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Aripiprazole | Olanzapine
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 7/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=15) | Olanzapine (N=15)
Akathisia (Psychiatric disorders) | 1 (1) | 7 (7) — Akathisia: mild or greater severity by subjective complaints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes